CLINICAL TRIAL: NCT02921659
Title: Safety & Efficacy of Nicotinamide Riboside Supplementation for Improving Physiological Function in Middle-Aged and Older Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: ChromaDex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0475
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Aging
Keywords: nicotinamide riboside; aging; arterial stiffness; endothelial dysfunction
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo, 500 mg, 2x/day for 6 weeks
  Interventions: Dietary Supplement: Placebo
- Niagen™ (Active Comparator): Niagen™ (nicotinamide riboside chloride, ChromaDex, Inc.) 500mg, 2x/day for 6 weeks.
  Interventions: Dietary Supplement: Niagen™

INTERVENTIONS:
Dietary Supplement: Niagen™ — nicotinamide riboside chloride, 250mg capsules
  Other Names: Nicotinamide Riboside
  Arms: Niagen™
Dietary Supplement: Placebo — silicified microcrystalline cellulose, vegetarian capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of supplementation with the Nicotinamide Adenine Dinucleotide (NAD+) precursor compound, Nicotinamide Riboside (NR), for improving physiological function (vascular, motor, and cognitive) in healthy middle-aged and older adults.

DETAILED DESCRIPTION:
Overall, the proposed research project has the long-term potential to influence clinical practice by establishing novel therapies for treating multiple domains of age-associated physiological dysfunction and thereby reducing the risk of clinical disease and disability.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Baseline brachial flow-mediated dilation (FMD) < 6%Δ (rationale: non-invasive screening to ensure exclusion of subjects with exceptionally high baseline endothelial function.
* Ability to perform motor and cognitive tests (e.g., can rise from a chair, walk for 2 min, climb 10 stairs)
* Women will be confirmed as postmenopausal (either natural or surgical) based on cessation of menses for >1 year.

Exclusion Criteria:

* ages <55 years or ≥80 years
* body mass index (BMI) >40 kg/m2 (rationale: vascular function and blood pressure measurements can be inaccurate in severely obese subjects and these subjects may differ in many ways from normal weight, overweight or less obese subjects)
* not weight stable in the prior 3 months (>2 kg weight change) or unwilling to remain weight stable throughout study (rationale: recent weight change or weight loss can influence vascular function)
* having unstable angina, acute myocardial infarction, coronary angioplasty, or aorto-coronary bypass surgery as defined by the occurrence of an event, symptom, surgery, or change in medication and/or dosage within 3 months prior to enrollment
* having thyroid disease that is not controlled by medications or <3 month's use of a particular medication and/or dosage (rationale: uncontrolled thyroid diseases are associated with alterations in vascular function)
* having past or present alcohol dependence or abuse, as defined by the American Psychiatry Association, Diagnostic and Statistical Manual of Mental Disorders
* abnormal blood chemistries for renal and liver function (>1 standard deviation outside the normal range)
* Moderate or severe peripheral artery disease (ankle-brachial index <0.7).
* Insufficient health to participate in a VO2max test based on a physical examination and/or graded exercise test (this will be determined in accordance with stated contraindications for exercise testing provided by the American Heart Association).

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 6 weeks
  self reported side effects, vital signs, hematology, liver enzymes, markers of kidney function and blood chemistry

SECONDARY OUTCOMES:
Endothelium Dependent Dilation | 6 weeks
  Brachial Artery Flow-Mediated Dilation (FMD)
Arterial Stiffness | 6 weeks
  Aortic Pulse Wave Velocity (PWV)
Cognitive Function | 6 weeks
  NIH Toolbox Cognitive Function Battery
Motor Function | 6 weeks
  NIH Toolbox Motor Function Battery
Systemic markers of oxidative stress and inflammation | 6 weeks
  Assessment of plasma C-reactive protein (CRP) and circulating and mononuclear cell-derived cytokine and antioxidant expression.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Martens, Ph.D., Principal Investigator — University of Colorado, Boulder
Locations (1):
- Clinical Translational Research Center, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description of Research Laboratory — http://www.colorado.edu/intphys/research/cardiovascular.html